CLINICAL TRIAL: NCT04285892
Title: Trial Investigating the Developmental Potential of Embryos Obtained After Biphasic in Vitro Oocyte Maturation (IVM) of Oocytes Including a Pre Maturation Culture Step ('capacitation Step') Compared with Standard IVM.
Brief Title: Embryo Developmental Potential in a Novel 2-step IVM System
Acronym: CAPA-IVM-Sib
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-CAPA-IVM-Sibling
Record Dates: First submitted 2020-02-14; First posted 2020-02-26 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: In Vitro Maturation of Oocytes

STUDY DESIGN:
Intervention Model Description: prospective randomized control trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CAPA IVM (Experimental): CAPA IVM is a 2-step In vitro Maturation system in which an additional culture step, in which the oocytes are kept in meiotic arrest by the presence of the C-type Natriuretic peptide (CNP) for 22-24 hours, is preceding the in vitro maturation step in which maturation medium is supplemented with amphiregulin (AREG). The 'IVM System' of Medicult-Origio is used as a base medium.
  Interventions: Device: CAPA-IVM
- Standard IVM (No Intervention): The IVM is performed as a single step protocol in which oocytes are immediately exposed to in vitro maturation medium for 30 hours. This is the current standard procedure in the clinical practice using the commercially available 'IVM System' of Medicult-Origio. Standard IVM medium: 10% HSA + 75mIU/ml FSH + 100mIU/ml hCG

INTERVENTIONS:
Device: CAPA-IVM — CAPA medium keeps oocytes in meiotic arrest for 22-24 hours. IVM medium allows oocytes to resume meiosis.
  CAPA medium: 10% human serum albumin (HSA) + 10nM estradiol (E2) + 25nM CNP + 5ng/ml Insulin + 1mIU/ml follicle stimulating hormone (FSH) IVM medium: 10% HSA + 10nM E2 + 5ng/ml Insulin + 101mIU/ml FSH + 100ng/ml AREG CNP: peptide naturally occurring in follicles to maintain meiotic arrest, E2: estrogen, enhances effects of CNP, Insulin: basic growth factor used in cell cultures and component of commercially available LAG medium of the standard IVM system, AREG: downstream effector of the LHCG receptor which helps meiotic resumption. HSA, FSH and hCG are CE labeled. CAPA IVM medium is currently not yet available as CE marked commercially available medium and needs to be prepared in house.
  Arms: CAPA IVM

SUMMARY:
In vitro maturation is a valid option for PCO(S) patients in the daily ART clinic, however maturation and embryologic development are not yet matching the efficiency levels obtained by standard COS treatment. To further enhance embryo quality after IVM, it was hypothesized to keep the connection and communication between oocyte and cumulus cells intact for a prolonged pre-maturation culture before IVM was initiated. This has been investigated and established using a meiotic blocker C-type Natriuretic peptide (CNP).

The CNP peptide is present in high concentrations in the growing follicle, is produced by the mural granulosa cell compartment and binds to the Natriuretic peptide receptor 2 (NRP2) present in the cumulus cells. Binding of CNP on NRP2 leads to intracellular cGMP increase in cumulus cells, which travels through the transzonal projections to the oocyte. In the oocyte, cGMP will block the resumption of meiosis.

Using CNP as natural inhibitor of meiosis, a new medium was designed to allow oocyte and surrounding cumulus cells to communicate and hence gain in competence for an additional culture period: the pre-maturation phase or Capacitation phase (CAPA). This system was devel-oped in mouse, tested in human in UZ Brussel on research material (toelating federaal EC: CFE-FCE ADV_073_ZUBrussel, toelating lokaal EC: 2016/411 BUN 143201630723) and used in a clinical setting in Vietnam.

DETAILED DESCRIPTION:
The current IVM system in use in the clinic has a single step approach and seems to be less efficient compared to research and literature findings using a biphasic CAPA-IVM system in terms of maturation.

To ascertain the efficiency of the biphasic CAPA-IVM system, both standard IVM and CAPA-IVM will be performed on sibling oocytes: maturation in standard IVM in the investigator's center is on average 47.5%, where CAPA-IVM reaches 62% maturation in literature.

The investigators aim to prove superiority of the CAPA-IVM system in terms of maturation. Also fertilization and embryo development will be compared.

The participants admitted to the study will be receiving both the standard IVM treatment for part of the participant's oocytes and the biphasic CAPA IVM system for the second part of the participant's oocytes.

In one ovary a regular oocyte pick up (OPU) will take place with oocytes assigned to the standard IVM treatment, in the other ovary the CAPA IVM system will be applied. This means oocytes that are liberated from the follicular environment need to be exposed immediately to the inhibiting CNP peptide and herefore the tubes to collect the follicle fluid from the punctured follicles are prefilled with CNP supplemented medium. The OPU procedure is identical for both ovaries and according to our standard OPU IVM procedure with the sole difference of empty or prefilled tubes to collect follicle fluid.

Oocytes from the 2 ovaries are separately processed in the lab according to attributed protocol.

After IVM of oocytes, mature oocytes are subjected to ICSI with partner's sperm or donor sperm. Partner's sperm sample will be frozen at the latest the day of egg retrieval and will be thawed the day of intracytoplasmic sperm injection (ICSI): due to the use of 2 different IVM protocols with 2 different time lines (30 hours maturation versus 24 hours+30 hours maturation), ICSI will take place on two consecutive days with a freshly thawed straw of sperm cells for each day.

Embryo development is followed until day 3 (cleavage stage) after ICSI. All embryos of sufficient quality will be vitrified for a deferred embryo transfer in a hormone replacement therapy (HRT) cycle. One embryo will be selected for embryo transfer based on the morphological quality assessment parameters, with the better quality as first choice for transfer, regardless the preceding IVM method. Frozen single embryo transfer cycles are repeated until pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* PCO(S) patients
* Anti-Mullerian Hormone ≥ 3.6 ng/mL
* Basal Antral Follicle Count ≥ 20
* All ranks of trial

Exclusion Criteria:

* Surgically obtained semen sample
* Grade 3 or 4 endometriosis, minor or major uterine abnormalities
* Preimplantation Genetic Testing
* Priming with Letrozole

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
oocyte maturation | oocyte maturation is assessed after 30 hours in the standard IVM protocol and after 54 hours after CAPA IVM
  the ability of the oocyte to extrude the first polar body

SECONDARY OUTCOMES:
Fertilization rate | The presence of 2 pronuclei is assessed between 18-20 hours after ICSI
  the ability of the oocyte to be activated and form pronuclei
morphologic parameters describing embryo quality per fertilized oocyte | embryo developmental assessment is performed 3 days after ICSI
  embryo developmental potential as estimated by morphological characteristics: embryos with 6 cells or more, less than 20% fragmentation, cell size according to the division pattern and the absence of multinucleated blastomeres are considered as good quality embryos. As secondary parameters, the presence of vacuoles or granulation in the majority of blastomeres will exclude the embryo from the 'good quality' group regardless of the earlier mentioned parameters.
utilization rate | utilization rate will be established 3 days after ICSI
  the embryos of sufficient quality to be vitrified for a deferred embryo transfer
embryo cryotolerance | First warming is done within one month after OPU in a new HRT cycle and repeated untill pregnancy up to 1 year after egg retrieval.
  the damage brought by the vitrification and warming process on cell survival within the embryo and the capacity of the vitrified/warmed embryo to resume cleavage divisions

CONTACTS AND LOCATIONS:
Overall Officials: Michel De Vos, MD, PhD, Principal Investigator — VUB- UZ Brussel
Locations (1):
- UZ Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saenz-de-Juano MD, Ivanova E, Romero S, Lolicato F, Sanchez F, Van Ranst H, Krueger F, Segonds-Pichon A, De Vos M, Andrews S, Smitz J, Kelsey G, Anckaert E. DNA methylation and mRNA expression of imprinted genes in blastocysts derived from an improved in vitro maturation method for oocytes from small antral follicles in polycystic ovary syndrome patients. Hum Reprod. 2019 Sep 29;34(9):1640-1649. doi: 10.1093/humrep/dez121. PMID 31398248
- [Background] Sanchez F, Le AH, Ho VNA, Romero S, Van Ranst H, De Vos M, Gilchrist RB, Ho TM, Vuong LN, Smitz J. Biphasic in vitro maturation (CAPA-IVM) specifically improves the developmental capacity of oocytes from small antral follicles. J Assist Reprod Genet. 2019 Oct;36(10):2135-2144. doi: 10.1007/s10815-019-01551-5. Epub 2019 Aug 9. PMID 31399916
- [Background] Vuong LN, Le AH, Ho VNA, Pham TD, Sanchez F, Romero S, De Vos M, Ho TM, Gilchrist RB, Smitz J. Live births after oocyte in vitro maturation with a prematuration step in women with polycystic ovary syndrome. J Assist Reprod Genet. 2020 Feb;37(2):347-357. doi: 10.1007/s10815-019-01677-6. Epub 2020 Jan 4. PMID 31902102
- [Background] Romero S, Sanchez F, Lolicato F, Van Ranst H, Smitz J. Immature Oocytes from Unprimed Juvenile Mice Become a Valuable Source for Embryo Production When Using C-Type Natriuretic Peptide as Essential Component of Culture Medium. Biol Reprod. 2016 Sep;95(3):64. doi: 10.1095/biolreprod.116.139808. Epub 2016 Aug 3. PMID 27488026
- [Background] Sanchez F, Lolicato F, Romero S, De Vos M, Van Ranst H, Verheyen G, Anckaert E, Smitz JEJ. An improved IVM method for cumulus-oocyte complexes from small follicles in polycystic ovary syndrome patients enhances oocyte competence and embryo yield. Hum Reprod. 2017 Oct 1;32(10):2056-2068. doi: 10.1093/humrep/dex262. PMID 28938744